CLINICAL TRIAL: NCT02423720
Title: Being Present: Audio-Based Mindfulness Meditation Intervention for Colorectal Cancer Patients and Caregivers
Brief Title: Mindfulness Meditation Intervention for Colorectal Cancer Patients and Caregivers
Acronym: Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15455
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Intervention (Other): Audio-based mindfulness intervention A 8-week single arm pilot study will be conducted among Helen Diller Famiily Comprehensive Cancer Center (HDFCCC) patients with metastatic colorectal cancer receiving chemotherapy and their caregivers (44 participants, total). Participants will receive an informational booklet containing a practice log and an MP3 player containing an introductory lecture and guided meditations. Practice reminders will be sent via text messages. Weekly emails will contain practice instructions and links to validated questionnaires.
  Interventions: Behavioral: Audio-Based Mindfulness

INTERVENTIONS:
Behavioral: Audio-Based Mindfulness — Audio-based mindfulness tracks (MP3 format).

SUMMARY:
This is a audio based mindfulness meditation intervention for colorectal cancer patients and caregivers. A 8-week single arm study will be conducted among University of California, San Francisco (UCSF) patients with metastatic colorectal cancer undergoing chemotherapy and caregivers of these patients (44 participants total).

DETAILED DESCRIPTION:
A metastatic cancer diagnosis is associated with high levels of distress in both patients and caregivers. The investigators hypothesize that an audio-based mindfulness intervention will be an effective means to reduce distress and improve quality of life among patients with advanced cancer and their caregivers. With the Being Present study, conduct an 8-week single arm study among UCSF patients with metastatic colorectal cancer undergoing chemotherapy and caregivers of these patients (44 participants total). Participants will receive an informational booklet containing a practice log and a MP3 player containing an introductory lecture and guided meditations. Practice reminders will be sent via text messages. Emails will contain practice assignments and links to validated survey instruments. The survey instruments (National Comprehensive Cancer Network (NCCN) Distress Thermometer and National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) adult short forms) will measure global health, anxiety, depression, fatigue, and sleep quality before, during, and after the intervention to obtain preliminary estimates of the efficacy of the intervention among patients and caregivers on self-reported outcomes. Qualitative data will be collected from pre- and post-intervention interviews.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must:

* Carry a diagnosis of metastatic colon, rectum, or small bowel adenocarcinoma
* Anticipate receiving chemotherapy for at least 12 weeks total from the time of recruitment
* Have life expectancy of at least 6 months
* Have Karnofsky Performance Status ≥60
* Be able to speak and read English
* Have access to a mobile phone
* Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet
* Have a distress level of ≥3 on the NCCN Distress Thermometer (DT).[1, 40]
* An effort will always be made to recruit patient and caregiver pairs, but unpaired patients are also eligible

Eligible caregivers are a spouse/partner, other family member, or a close friend of a patient with metastatic colon, rectum, or small bowel adenocarcinoma.

Eligible caregivers must:

* Be able to speak and read English
* Have access to a mobile phone
* Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet

Exclusion Criteria:

This study is limited the study to patients with metastatic colon, rectum, or small bowel adenocarcinoma, because treatment regimens and disease trajectories for these disease groups are similar.

Deafness, Current meditation practice (>2 episodes or >1 hour total, weekly), and current enrollment in a stress reduction program are exclusion criteria for the intervention study because the study is designed as an audio-based introduction to mindfulness meditation.

Patients with a DT level >7 will be considered on a case-by- case basis. Patients and caregivers who participate in a focus group and meet criteria for the intervention will be given the opportunity to participate: data will be collected, but these patients/participants will not be included in the final analyses so as not to bias the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible patients and caregivers who agree to be screened, consent to participate, and complete or partially complete the intervention, as a measure of feasibility and acceptability. | 8 weeks
Adherence to the intervention, as assessed by frequency and duration of practicing the exercises (recorded in a log and responses to text messages) | 8 weeks

SECONDARY OUTCOMES:
Reasons for ineligibility, as a measure of feasibility | 8 weeks
Proportion of enrolled patients and caregivers who refuse to participate in or complete the intervention, as a measure of feasibility and acceptability | 8 weeks
Reasons for non-participation/non-continuation of the intervention, as a measure of feasibility and acceptability | 8 weeks
Adherence to the intervention, as assessed by frequency and duration of practicing the exercises (recorded in a log and responses to text messages) | 8 weeks

OTHER OUTCOMES:
Quality of life, as assessed by NIH PROMIS instruments at the beginning, midpoint and end of the study | 0, 4 and 8 weeks
Distress, as assessed by NCCN Distress Thermometer and NIH PROMIS instruments at the beginning, midpoint and end of the study | 0, 4 and 8 weeks
Anxiety, as assessed by NCCN Distress Thermometer and NIH PROMIS instruments at the beginning, midpoint and end of the study | 0, 4 and 8 weeks
Depression, as assessed by NCCN Distress Thermometer and NIH PROMIS instruments at the beginning, midpoint and end of the study | 0, 4 and 8 weeks
Fatigue, as assessed by NCCN Distress Thermometer and NIH PROMIS instruments at the beginning, midpoint and end of the study | 0, 4 and 8 weeks
Sleep quality, as assessed by NCCN Distress Thermometer and NIH PROMIS instruments at the beginning, midpoint and end of the study | 0, 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Atreya, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Atreya CE, Kubo A, Borno HT, Rosenthal B, Campanella M, Rettger JP, Joseph G, Allen IE, Venook AP, Altschuler A, Dhruva A. Being Present: A single-arm feasibility study of audio-based mindfulness meditation for colorectal cancer patients and caregivers. PLoS One. 2018 Jul 23;13(7):e0199423. doi: 10.1371/journal.pone.0199423. eCollection 2018. PMID 30036361